CLINICAL TRIAL: NCT03753165
Title: Effect of High Intensity Interval Exercise on Pain,Disability, and Autonomic Nervous System on Chronic Low Back Pain Patients
Brief Title: Effect of High Intensity Interval Exercise on Chronic Low Back Pain Patients
Acronym: CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Haya Mohammad ALMaawi, Principal Investigator, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-PGS-2018-01-076
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain, Heart rate variability
MeSH Terms: interventions — High-Intensity Interval Training; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: It is a single blinded randomised clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Exercise group (Experimental): Patients suffering from chronic low back pain perform 12 sessions of high intensity interval exercise (HIIE) over a period of 6 weeks at an intensity of 80% of their maximal Heart rate. In addition they also receive conventional physiotherapy in the form of hot pack or TENS
  Interventions: Other: High intensity interval exercise
- Conventional physiotherapy (No Intervention): Patients suffering from chronic low back pain will receive conventional physiotherapy such as TENS and hot packs applied over appropriate areas over a period of 6 weeks

INTERVENTIONS:
Other: High intensity interval exercise — High intensity interval exercise at 80% of the maximal heart rate derived from the maximal graded exercise. Each individual will undergo 12 sessions of HIIE over a period of six weeks
  Other Names: Conventional physiotherapy- Hot packs, TENS
  Arms: High Intensity Interval Exercise group

SUMMARY:
Patients with low back pain (LBP) often report an overall reduced physical activity and fitness that could consequently lead to an altered autonomic balance. Dysregulation of autonomic nervous system (ANS) is also implicated to be an underlying cause in the initiation and persistence of chronic muscle pain.High intensity interval exercise (HIIE) is a newer modality where short bursts of high intensity exercise are interspersed with rest intervals.

Method:Study Design: It is a single blinded randomised clinical trial.Sample Size:

Experimental Group (HIIE+ standard regular physiotherapy) = 40 Positive Control Group (standard regular physiotherapy) = 40 After the ethical approval of Imam Abdulrahman Bin Faisal University, Dammam, eighty (80) patients with nonspecific CLBP (either sex, age range 18-65 years years) will be recruited. These patients, with mild to moderate disability/pain according to Oswestry index, will be referred from the orthopedics clinic, rheumatologist, neurology, rehabilitation specialist, to the physiotherapy department.

Oswestry Disability Index (ODI) will be completed for all CLBP patients. Pre and post assessment includes pain intensity, disability, resting heart rate (HRrest) and blood pressure, maximum heart rate (HRmax) after graded maximal exercise, heart rate recovery after graded maximal exercise (HRR).

Tests of autonomic function will be done by recording ECG and analyzing he ECG for variability in heart rate (HRV), the Expiratory/inspiratory ratio in deep breathing (HRVdb) and baroreceptor sensitivity (BRS) at rest. Additionally each subject will be exposed to an orthostatic challenge and his responses will be evaluated. The recording will be done first in supine position and then asking the patient to quickly stand up and remain standing for 5 min. Data will be entered in Microsoft excel and comparisons and correlations will be done using either excel or SPSS version 20.

DETAILED DESCRIPTION:
Effect of High Intensity Interval Exercise on pain, disability and autonomic balance in patients with chronic low back pain

Chronic low back pain (CLBP) is a clinical problem of large magnitude with great socio-economical effect. About 80% of people may complain of low back pain in their life.

Patients with low back pain (LBP) often report an overall reduced physical activity and fitness that could consequently lead to an altered autonomic balance. Dysregulation of autonomic nervous system (ANS) is also implicated to be an underlying cause in the initiation and persistence of chronic muscle pain. Different types of exercises can be prescribed to patients with CLBP to improve pain, disability and physical fitness. High intensity interval exercise (HIIE) is a newer modality where short bursts of high intensity exercise are interspersed with rest intervals.it is more time efficient, enjoyable, and superior to mild or moderate intensity continuous exercise in improving the physical fitness, peak performance, autonomic balance, muscle strength and coordination in athletes. HIIE might prove more useful and effective for individuals with nonspecific CLBP and could have a better adherence rate in the long run.

Methods: After the ethical approval of Imam Abdulrahman Bin Faisal University, Dammam, KSA, eighty (80) patients with nonspecific CLBP (either sex, age: 18-65 years) will be recruited. These patients, with mild to moderate disability/pain according to Oswestry index, will be referred from relevant clinics to the physiotherapy department of King Fahd Hospital of the University, AlKhobar (KFHU). After full explanation of the study, the patients will be required to sign an informed consent form and then they will be randomly assigned to one of the two groups.

Experimental Group (GE: n= 40) will be assigned for HIIE in addition to standard regular physiotherapy, and Control Group (GC: n=40) will be designated as control group with standard regular physiotherapy only. Pre and post intervention assessment includes pain intensity through Numerical Pain Scale, disability through Oswestry Disability Index (ODI) and autonomic balance through heart rate variability (HRV) and baroreflex sensitivity (BRS) at rest and in response to an orthostatic challenge.

Data will be entered in Microsoft excel and comparisons and correlations will be done using either excel or SPSS version 20 Expectations: It is expected that HIIE will improve the autonomic balance of the CLBP patients to a greater extent compared to no-exercise and consequently improve the pain and disability to a higher degree. HIIE could be a useful, efficacious addition to the list of exercise modalities for patients with nonspecific CLBP, and could be recommended for management of appropriate group of CLBP patients.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-65 years.
* BMI 18.5 - 34.9 kg/m2.
* Diagnosed patients as non-specific chronic low back pain patients, referred by orthopedic specialist, rheumatologist, rehabilitation specialist to physical therapy.
* Oswestry Disability Index (ODI): mild to moderate .
* The subjects should be able to understand, communicate and perform the examination and can walk without any walking aids.

Exclusion Criteria:

* Walking with using any walking aids.
* Subjects with secondary LBP, Sciatica, Osteoporosis, Osteoarthritis, generalized neuromuscular problem or any deformity.
* Any diagnosed disease likely to interfere with exercise on bicycle ergometer or safety of the subject (especially cardiac or respiratory disease.
* Patients with known diabetic autonomic complications
* Persons taking medicines that are known to interfere with HRV variables, such as beta blockers, calcium antagonists.
* Pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability | baseline and 6 weeks
  heart rate variability parameters including SDNN, RMSSD, LF, HF, LH/HF

SECONDARY OUTCOMES:
Heart Rate Recovery | baseline and after 6 weeks
  Heart rate recovery from the peak rate at 1st, 2nd and 3rd minute after cessation of heavy exercise
Numerical pain scale | baseline and after 6 weeks
  Measurement of pain intensity
Oswestry Disability Index | baseline and after 6 weeks
  Questionnaire to assess the disability in patients with chronic low back pain
Baroreceptor Sensitivity (BRS) | baseline and 6 weeks
  recording of finger arterial blood pressure and interbeat interval with finometer and calculating the baroreceptor sensitivity with dedicated software PRVBRS

CONTACTS AND LOCATIONS:
Locations (1):
- King Fahd Hospital of the University, Khobar, Eastren, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
No there is no plan to make the IPD available

REFERENCES:
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. J Pain. 2014 Jun;15(6):569-85. doi: 10.1016/j.jpain.2014.03.005. Epub 2014 Apr 29. PMID 24787228
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle: Part I: cardiopulmonary emphasis. Sports Med. 2013 May;43(5):313-38. doi: 10.1007/s40279-013-0029-x. PMID 23539308
- [Background] Cole CR, Blackstone EH, Pashkow FJ, Snader CE, Lauer MS. Heart-rate recovery immediately after exercise as a predictor of mortality. N Engl J Med. 1999 Oct 28;341(18):1351-7. doi: 10.1056/NEJM199910283411804. PMID 10536127
- [Background] Dupuy O, Mekary S, Berryman N, Bherer L, Audiffren M, Bosquet L. Reliability of heart rate measures used to assess post-exercise parasympathetic reactivation. Clin Physiol Funct Imaging. 2012 Jul;32(4):296-304. doi: 10.1111/j.1475-097X.2012.01125.x. Epub 2012 Feb 23. PMID 22681607
- [Background] Fisher G, Brown AW, Bohan Brown MM, Alcorn A, Noles C, Winwood L, Resuehr H, George B, Jeansonne MM, Allison DB. High Intensity Interval- vs Moderate Intensity- Training for Improving Cardiometabolic Health in Overweight or Obese Males: A Randomized Controlled Trial. PLoS One. 2015 Oct 21;10(10):e0138853. doi: 10.1371/journal.pone.0138853. eCollection 2015. PMID 26489022
- [Background] Fairbank J. Use of Oswestry Disability Index (ODI). Spine (Phila Pa 1976). 1995 Jul 1;20(13):1535-7. No abstract available. PMID 8623078
- [Background] Fletcher GF, Ades PA, Kligfield P, Arena R, Balady GJ, Bittner VA, Coke LA, Fleg JL, Forman DE, Gerber TC, Gulati M, Madan K, Rhodes J, Thompson PD, Williams MA; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Nutrition, Physical Activity and Metabolism, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation. 2013 Aug 20;128(8):873-934. doi: 10.1161/CIR.0b013e31829b5b44. Epub 2013 Jul 22. No abstract available. PMID 23877260
- [Background] Freeman R, Chapleau MW. Testing the autonomic nervous system. Handb Clin Neurol. 2013;115:115-36. doi: 10.1016/B978-0-444-52902-2.00007-2. PMID 23931777
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] Hallman DM, Ekman AH, Lyskov E. Changes in physical activity and heart rate variability in chronic neck-shoulder pain: monitoring during work and leisure time. Int Arch Occup Environ Health. 2014;87(7):735-44. doi: 10.1007/s00420-013-0917-2. Epub 2013 Oct 26. PMID 24162088
- [Background] Iellamo F, Manzi V, Caminiti G, Sposato B, Massaro M, Cerrito A, Rosano G, Volterrani M. Dose-response relationship of baroreflex sensitivity and heart rate variability to individually-tailored exercise training in patients with heart failure. Int J Cardiol. 2013 Jun 20;166(2):334-9. doi: 10.1016/j.ijcard.2011.10.082. Epub 2011 Nov 9. PMID 22078985
- [Background] Jung ME, Bourne JE, Beauchamp MR, Robinson E, Little JP. High-intensity interval training as an efficacious alternative to moderate-intensity continuous training for adults with prediabetes. J Diabetes Res. 2015;2015:191595. doi: 10.1155/2015/191595. Epub 2015 Mar 30. PMID 25918728
- [Background] La Rovere MT, Pinna GD, Maestri R, Sleight P. Clinical value of baroreflex sensitivity. Neth Heart J. 2013 Feb;21(2):61-3. doi: 10.1007/s12471-012-0349-8. PMID 23184601
- [Background] Perini R, Veicsteinas A. Heart rate variability and autonomic activity at rest and during exercise in various physiological conditions. Eur J Appl Physiol. 2003 Oct;90(3-4):317-25. doi: 10.1007/s00421-003-0953-9. Epub 2003 Sep 12. PMID 13680241
- [Background] Pinna GD, Maestri R, La Rovere MT. Assessment of baroreflex sensitivity from spontaneous oscillations of blood pressure and heart rate: proven clinical value? Physiol Meas. 2015 Apr;36(4):741-53. doi: 10.1088/0967-3334/36/4/741. Epub 2015 Mar 23. PMID 25798657